CLINICAL TRIAL: NCT02122666
Title: Modulating Physiologic Effects Of Phospholipid Metabolism In Obesity And Diabetes; AIM 4: Composition and Function of Sarcoplasmic Reticulum in Persons With the Metabolic Syndrome
Brief Title: Composition & Function of Sarcoplasmic Reticulum in Persons With the Metabolic Syndrome
Acronym: COMP-SR
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: HRPO201311099
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Pre-diabetes; impaired glucose tolerance; Phospholipids
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and frozen tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metabolic Syndrome: Muscle biopsy to determine sarcoplasmic reticulum composition and function, Oral Glucose tolerance test with insulin levels at time points to determine Insulin sensitivity, DEXA scan to determine lean muscle and fat mass
  Interventions: Procedure: muscle biopsy
- Control: Muscle biopsy to determine sarcoplasmic reticulum composition and function, Oral Glucose tolerance test with insulin levels at time points to determine Insulin sensitivity, DEXA scan to determine lean muscle and fat mass
  Interventions: Procedure: muscle biopsy

INTERVENTIONS:
Procedure: muscle biopsy — A member of the study team will obtain a small sample of muscle tissue from the patient's thigh (vastus lateralis muscle).

SUMMARY:
The investigators previous research has suggested that lipid (fatty) composition in the muscle cells of mice plays a key role in their insulin sensitivity. The purpose of this study is to determine whether these specific fat signatures translate to humans by comparing the muscle of healthy patients to those with pre-diabetes, or "the metabolic syndrome".

DETAILED DESCRIPTION:
The Comp-SR study explores the role of lipid metabolism in key metabolic pathways in skeletal muscle. It is a translation of previous research done in mice studying the effects and functions of certain key enzymes involved in lipid metabolism found to be associated with insulin resistance. These enzymes are fatty acid synthase (FAS), choline/ethanolamine phosphotransferase 1 (CEPT1) and sarcoplasmic-endoplasmic reticulum ATPase (SERCA). Based on the investigators research, it appears that the activity and function of these enzymes determines the ratio of certain phospholipids in the sarcoplasmic reticulum (SR), namely phosphatidylethanolamine (PE) and phosphatidylcholine (PC). Furthermore, the investigators have found that the ratio of these phospholipids correlates with the mouse's sensitivity to insulin.

Based on the muscle biopsies of four healthy persons, it was found that human muscle contains similar phospholipids and phospholipid ratios to mice. It is hypothesized that these phospholipid signatures may be predictive of the metabolic status of humans as well. The specific aims of this study are to determine if the composition and function of the sarcoplasmic reticulum is altered in persons with the metabolic syndrome compared to lean controls. This knowledge could provide new understanding of impediments to effective therapy, novel biomarkers of disease progression, and innovative treatment targets for diabetes.

ELIGIBILITY:
Control subjects

Inclusion:

Sedentary: No routine exercise, walking <10,000 steps per day Age >18 and <65 Body Mass Index (BMI) <32 Healthy by physical exam (patient is devoid of major acute or chronic illness) No significant abnormality in screening labs

Exclusion:

Currently on any significant prescription medications other than oral contraceptives in women Currently Pregnant Current Tobacco Use

Subjects with the Metabolic Syndrome

Inclusion:

Sedentary: No routine exercise, walking <10,000 steps per day Age >18 and <65 Body Mass Index (BMI) >30

Meet at least three of the following Adult Treatment Panel (ATP) III criteria for the metabolic syndrome:

waist circumference > or = 40 inches in men, > or = 35 inches in women blood triglycerides > or = 150 mg/dL blood HDL cholesterol <40 mg/dL in men, <50 in women blood pressure > or = 130 mmHg systolic, or > or = 85 mmHg diastolic fasting blood sugar > or = 100 mg/dL

Exclusion:

Diagnosed with Type 2 diabetes, coronary artery disease, cancer, liver, lung, or kidney disease or any other major illness

Currently on any significant prescription medications other than:

oral contraceptives in women More than two standard medication for stage 1 hypertension in men or women (blood pressure 140-159/90-99) Currently Pregnant Current Tobacco Use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-03; Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay F. Semenkovich, M.D., Principal Investigator — Washington University School of Medicine; Janet B McGill, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Finucane MM, Stevens GA, Cowan MJ, Danaei G, Lin JK, Paciorek CJ, Singh GM, Gutierrez HR, Lu Y, Bahalim AN, Farzadfar F, Riley LM, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Body Mass Index). National, regional, and global trends in body-mass index since 1980: systematic analysis of health examination surveys and epidemiological studies with 960 country-years and 9.1 million participants. Lancet. 2011 Feb 12;377(9765):557-67. doi: 10.1016/S0140-6736(10)62037-5. Epub 2011 Feb 3. PMID 21295846
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Regensteiner JG, Sippel J, McFarling ET, Wolfel EE, Hiatt WR. Effects of non-insulin-dependent diabetes on oxygen consumption during treadmill exercise. Med Sci Sports Exerc. 1995 Jun;27(6):875-81. PMID 7658949
- [Background] Funai K, Song H, Yin L, Lodhi IJ, Wei X, Yoshino J, Coleman T, Semenkovich CF. Muscle lipogenesis balances insulin sensitivity and strength through calcium signaling. J Clin Invest. 2013 Mar;123(3):1229-40. doi: 10.1172/JCI65726. Epub 2013 Feb 8. PMID 23376793
- [Background] McGarry JD. What if Minkowski had been ageusic? An alternative angle on diabetes. Science. 1992 Oct 30;258(5083):766-70. doi: 10.1126/science.1439783.
- [Background] Kiens B. Skeletal muscle lipid metabolism in exercise and insulin resistance. Physiol Rev. 2006 Jan;86(1):205-43. doi: 10.1152/physrev.00023.2004. PMID 16371598
- See also: Washington U in St. Louis, Endocrinology Current Clinical Studies — http://endo.wustl.edu/current-clinical-studies/
- See also: Clay F. Semenkovich, MD — http://endo.wustl.edu/clay-f-semenkovich-m-d/
- See also: Washington U in St. Louis; Research Participant Registry — https://vfh.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metabolic Syndrome | Control
Started | 12 | 15
Completed | 12 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metabolic Syndrome | Control | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (8.4) | 39.5 (16.4) | 44.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sarcoplasmic Reticulum Composition
Description: We will take a muscle tissue sample from the subject's thigh (vastus lateralis) to quantify phosphatidylcholine to phosphatidylethanolamine ratio of the sarcoplasmic reticulum.
Time Frame: Study Visit Week 4
Population: Samples not included were lost during tissue processing. Metabolic syndrome (n=10); Control (n=13)
Measure: Mean (Standard Error); unit: PC:PE ratio
Arm/Group | Metabolic Syndrome | Control
Number analyzed (Participants) | 10 | 13
PC:PE ratio | 2.0 (0.2) | 2.2 (0.2)

2. Secondary Outcome: Insulin Sensitivity
Description: The homeostatic model assessment for insulin resistance (HOMA-IR) is a calculated value using fasting glucose and insulin levels. It provides a measure of insulin resistance. HOMA-IR values between 0.5 and 1.4 are considered normal and values >2.9 indicate insulin resistance. The Matsuda Index reflects insulin sensitivity. It is calculated from glucose and insulin levels drawn fasting and during an OGTT. Matsuda Index values of 2.5 or higher are normal and indicate lack of insulin resistance or normal insulin sensitivity. Results of these measures are displayed graphically in the published paper.
Time Frame: Study visit week 4
Population: Oral glucose tolerance tests were performed on 15 controls and 11 metabolic syndrome participants. The insulin data was lost for one metabolic syndrome participant.
Measure: Mean (Standard Deviation); unit: Matsuda Index
Arm/Group | Metabolic Syndrome | Control
Number analyzed (Participants) | 11 | 15
Matsuda Index | 2.5 (1.9) | 5.6 (2.2)

3. Secondary Outcome: Lean and Fat Body Mass
Description: We will perform a Duel Energy X-ray absorptiometry (DEXA) scan to approximate lean and fat body mass of study subjects.
Time Frame: Study Visit week 4
Population: All study participants received DEXAs and data were reported.
Measure: Mean (Standard Deviation); unit: Total body fat (%)
Arm/Group | Metabolic Syndrome | Control
Number analyzed (Participants) | 12 | 15
Total body fat (%) | 43.7 (5.0) | 30.6 (7.5)

ADVERSE EVENTS:
Time Frame: Individual study participation: 4-6 weeks Study duration of entire cohort: 9 years, 11 months
Description: Our definition of adverse / serious adverse events do not differ from clinicaltrials.gov.
Arm/Group | Metabolic Syndrome | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02122666/Prot_SAP_000.pdf